CLINICAL TRIAL: NCT01498705
Title: The Natural History of Procalcitonin in Hemorrhagic Stroke
Status: Withdrawn | Type: Observational
Why Stopped: Anticipated grant was withdrawn and additional funding was unable to be obtained
Sponsor: CAMC Health System (Other)
Responsible Party: Principal Investigator, Carol Morreale, Clinical Pharmacist Specialist, CAMC Health System
Other Study IDs: 1997096
Record Dates: First submitted 2011-12-20; First posted 2011-12-23 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Intraventricular Hemorrhage; Intracerebral Hemorrhage
Keywords: Intraventricular Hemorrhage; Intracerebral Hemorrhage; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Procalcitonin Level
MeSH Terms: conditions — Cerebral Hemorrhage; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases | interventions — Procalcitonin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 3 mL of blood will be obtained for each PCT sample and will be sent to the Virology lab at CAMC Memorial hospital where the serum will be frozen until all samples are collected. After all samples from each of the 30 patients are obtained, the specimens will be analyzed for the PCT value and then discarded.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemmorhagic Stroke: * Hospitalization for an admitting diagnosis of hemorrhagic stroke admitted to the neurosurgical intensive care unit
  * Age greater than 18 years
  * No evidence of ischemic cerebrovascular injury
  Interventions: Other: Procalcitonin level

INTERVENTIONS:
Other: Procalcitonin level — PCT level upon admission and on days 1, 3, and 5 following baseline level

SUMMARY:
Approximately 12% of strokes in the United States are hemorrhagic.1 Hemorrhagic stroke can lead to multiple complications including fever that is not infectious. Identifying the cause of fever can help physicians choose the best care for the patient to try and prevent further damage to the already injured brain. Bacterial infection is one possible cause of fever in the stroke patient; however an incorrect diagnosis of infection can lead to unnecessary antibiotic use. Better screening tools for infection are being developed to help fight the problem of antibiotic resistance and unnecessary antibiotic use. Unnecessary use of antibiotics in patients increases the risk of adverse events and overall healthcare costs. Procalcitonin (PCT) is one such screening tool which has been used previously to help tell apart bacterial and nonbacterial causes of infection in other disease states; however, PCT has not been studied in hemorrhagic stroke patients. The purpose of this study is to understand the progress of PCT in hemorrhagic stroke patients in order to see whether PCT can be a useful marker for infection in these patients.

DETAILED DESCRIPTION:
Stroke is the second leading killer worldwide and the third leading cause of death in the United States. The two major mechanisms causing brain damage in stroke are, ischemia and hemorrhage. Several complications can arise from these cerebral insults ranging from minor neurologic dysfunction, complete immobility, or death. In the intensive care setting, clinicians combat the pathophysiologic processes that lead to the aforementioned sequelae of stroke and contest other acute issues which may or may not be secondary to the stroke itself, with one such issue being hyperthermia. Hyperthermia is defined by the Society of Critical Care Medicine as a temperature greater than 38.3°C. In one prospective study, hyperthermia was reported to occur in 43% of patients during the first week of hospitalization following an ischemic or hemorrhagic (excluding subarachnoid hemorrhage) stroke. Hyperthermia in the stroke patient can be detrimental leading to increased infarct size and worsened neurological outcomes. The etiology of the hyperthermia may not be clear upon initial evaluation but cessation of fever is essential to prevent further damage.

One possible cause of hyperthermia in the stroke patient is bacterial infection. Infection complicating cerebral insult can lead to poor functional outcome and increased mortality. Kilpatrick and colleagues found that fever occurred in 47% of patients who were admitted with either a traumatic or ischemic brain injury and 70% of these patients received at least one antibiotic within 24 hours of their febrile episode, however the antibiotics had no effect on controlling the fevers. With bacterial resistance ever increasing, it is vital that clinicians reserve antibiotics for patients in whom the source of fever is believed to be secondary to an infectious process. It has been estimated that the United States health care system spends more than $20 billion annually on antibiotic-resistant infections and these infections result in more than eight million additional hospital days. Antibiotic use across health care disciplines has been estimated to be administered either inappropriately or unnecessarily 50% of the time. Considering clinical symptoms of infection can mirror other disease processes, reliable diagnostic biomarkers would be useful in helping determine the appropriate diagnosis.

PCT is a 116 amino acid peptide with a sequence identical to calcitonin but lacking hormonal activity. PCT was first utilized by Assicot et al in the setting of sepsis to help determine whether the inflammatory response from the patient was secondary to bacterial infection. Since this finding, PCT has been shown in several studies to have a high sensitivity and specificity for indicating systemic bacterial infections. During infection PCT is secreted into the bloodstream without increasing calcitonin. PCT has been shown prospectively to only be elevated in patients with bacterial infections while remaining consistently low in patients infected with viruses or other inflammatory processes. Often when insulted, the body utilizes proteins and metabolic products, and the changes noted in these substances are often used as markers of inflammation. Unlike erythryocyte sedimentation rate (ESR) and C-reactive protein (CRP), PCT remains low during these inflammatory states. Furthermore, it has been shown that PCT levels increase earlier after stimulation (3-6hrs) compared to C-reactive protein (12-24hrs), indicating PCT can be utilized to rapidly detect bacterial infections. Normal PCT levels in adults are less than 0.1 ng/mL while PCT values greater than 0.5ng/mL have been determined to be predictive of bacterial infection. PCT has been evaluated in several clinical scenarios to help determine a bacterial versus a non-bacterial source of infection, however, to our knowledge, the effects of hemorrhagic stroke on PCT are not yet known. Determining the natural history of PCT in a hemorrhagic stroke patient would provide beneficial information as to whether PCT can be used as a biomarker in this population to help differentiate a bacterial from a non-bacterial cause of hyperthermia.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for an admitting diagnosis of hemorrhagic stroke admitted to the neurosurgical intensive care unit
* Age greater than 18 years
* No evidence of ischemic cerebrovascular injury

Exclusion Criteria:

* Concomitant traumatic brain injury
* Antibiotics on admission to the NICU
* Immunocompromised by chemotherapy or HIV positive or patient with neutropenia (ANC <1000)
* Women who are pregnant and/or of childbearing age where a pregnancy test has not already occurred

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Neurosurgical ICU with a diagnosis of intraventricular or intracerebral hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Natural progression of PCT following hemorrhagic stroke | Change in serum PCT level on day 0 (baseline) from serum PCT level day 1, 3, and 5.

SECONDARY OUTCOMES:
Markers of infection (if obtained by treating medical team) using SIRS criteria well as cultures. | From date of enrollment to 28 days or until death or discharge, whichever comes first.
  Sirs criteria: temperature < 36°C or > 38°C, heart rate > 90 beats/min, respiratory rate > 20 breaths/min, white blood cell count < 4000/mm² or > 12,000/mm² or ≥ 10% bands Cultures: blood, urine and sputum obtained by the treating medical team during study period and followed until final culture results are determined

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W Haden, MD, Principal Investigator — WVU School of Medicine/Charleston Division
Locations (1):
- Charleston Area Medical Center, Charleston, West Virginia, United States

REFERENCES:
- [Background] Roberts RR, Hota B, Ahmad I, Scott RD 2nd, Foster SD, Abbasi F, Schabowski S, Kampe LM, Ciavarella GG, Supino M, Naples J, Cordell R, Levy SB, Weinstein RA. Hospital and societal costs of antimicrobial-resistant infections in a Chicago teaching hospital: implications for antibiotic stewardship. Clin Infect Dis. 2009 Oct 15;49(8):1175-84. doi: 10.1086/605630. PMID 19739972
- [Background] Meyer BC, Hemmen TM, Jackson CM, Lyden PD. Modified National Institutes of Health Stroke Scale for use in stroke clinical trials: prospective reliability and validity. Stroke. 2002 May;33(5):1261-6. doi: 10.1161/01.str.0000015625.87603.a7. PMID 11988601
- [Background] Castelli GP, Pognani C, Cita M, Paladini R. Procalcitonin as a prognostic and diagnostic tool for septic complications after major trauma. Crit Care Med. 2009 Jun;37(6):1845-9. doi: 10.1097/CCM.0b013e31819ffd5b. PMID 19384224
- [Result] O'Grady NP, Barie PS, Bartlett JG, Bleck T, Carroll K, Kalil AC, Linden P, Maki DG, Nierman D, Pasculle W, Masur H; American College of Critical Care Medicine; Infectious Diseases Society of America. Guidelines for evaluation of new fever in critically ill adult patients: 2008 update from the American College of Critical Care Medicine and the Infectious Diseases Society of America. Crit Care Med. 2008 Apr;36(4):1330-49. doi: 10.1097/CCM.0b013e318169eda9. PMID 18379262
- [Result] Azzimondi G, Bassein L, Nonino F, Fiorani L, Vignatelli L, Re G, D'Alessandro R. Fever in acute stroke worsens prognosis. A prospective study. Stroke. 1995 Nov;26(11):2040-3. doi: 10.1161/01.str.26.11.2040. PMID 7482646
- [Result] Dietrich WD, Alonso O, Halley M, Busto R. Delayed posttraumatic brain hyperthermia worsens outcome after fluid percussion brain injury: a light and electron microscopic study in rats. Neurosurgery. 1996 Mar;38(3):533-41; discussion 541. doi: 10.1097/00006123-199603000-00023. PMID 8837806
- [Result] Hong KS, Kang DW, Koo JS, Yu KH, Han MK, Cho YJ, Park JM, Bae HJ, Lee BC. Impact of neurological and medical complications on 3-month outcomes in acute ischaemic stroke. Eur J Neurol. 2008 Dec;15(12):1324-31. doi: 10.1111/j.1468-1331.2008.02310.x. PMID 19049549
- [Result] Katzan IL, Cebul RD, Husak SH, Dawson NV, Baker DW. The effect of pneumonia on mortality among patients hospitalized for acute stroke. Neurology. 2003 Feb 25;60(4):620-5. doi: 10.1212/01.wnl.0000046586.38284.60. PMID 12601102
- [Result] Johnston KC, Li JY, Lyden PD, Hanson SK, Feasby TE, Adams RJ, Faught RE Jr, Haley EC Jr. Medical and neurological complications of ischemic stroke: experience from the RANTTAS trial. RANTTAS Investigators. Stroke. 1998 Feb;29(2):447-53. doi: 10.1161/01.str.29.2.447. PMID 9472888
- [Result] Langhorne P, Stott DJ, Robertson L, MacDonald J, Jones L, McAlpine C, Dick F, Taylor GS, Murray G. Medical complications after stroke: a multicenter study. Stroke. 2000 Jun;31(6):1223-9. doi: 10.1161/01.str.31.6.1223. PMID 10835436
- [Result] Kilpatrick MM, Lowry DW, Firlik AD, Yonas H, Marion DW. Hyperthermia in the neurosurgical intensive care unit. Neurosurgery. 2000 Oct;47(4):850-5; discussion 855-6. doi: 10.1097/00006123-200010000-00011. PMID 11014424
- [Result] El-Solh AA, Vora H, Knight PR 3rd, Porhomayon J. Diagnostic use of serum procalcitonin levels in pulmonary aspiration syndromes. Crit Care Med. 2011 Jun;39(6):1251-6. doi: 10.1097/CCM.0b013e31820a942c. PMID 21283001
- [Result] Assicot M, Gendrel D, Carsin H, Raymond J, Guilbaud J, Bohuon C. High serum procalcitonin concentrations in patients with sepsis and infection. Lancet. 1993 Feb 27;341(8844):515-8. doi: 10.1016/0140-6736(93)90277-n. PMID 8094770
- [Result] Chalupa P, Beran O, Herwald H, Kasprikova N, Holub M. Evaluation of potential biomarkers for the discrimination of bacterial and viral infections. Infection. 2011 Oct;39(5):411-7. doi: 10.1007/s15010-011-0126-4. Epub 2011 Jul 1. PMID 21720792
- [Result] Hochreiter M, Kohler T, Schweiger AM, Keck FS, Bein B, von Spiegel T, Schroeder S. Procalcitonin to guide duration of antibiotic therapy in intensive care patients: a randomized prospective controlled trial. Crit Care. 2009;13(3):R83. doi: 10.1186/cc7903. Epub 2009 Jun 3. PMID 19493352
- [Result] Gendrel D, Bohuon C. Procalcitonin as a marker of bacterial infection. Pediatr Infect Dis J. 2000 Aug;19(8):679-87; quiz 688. doi: 10.1097/00006454-200008000-00001. No abstract available. PMID 10959733
- [Result] Adams HP Jr, del Zoppo G, Alberts MJ, Bhatt DL, Brass L, Furlan A, Grubb RL, Higashida RT, Jauch EC, Kidwell C, Lyden PD, Morgenstern LB, Qureshi AI, Rosenwasser RH, Scott PA, Wijdicks EF; American Heart Association; American Stroke Association Stroke Council; Clinical Cardiology Council; Cardiovascular Radiology and Intervention Council; Atherosclerotic Peripheral Vascular Disease and Quality of Care Outcomes in Research Interdisciplinary Working Groups. Guidelines for the early management of adults with ischemic stroke: a guideline from the American Heart Association/American Stroke Association Stroke Council, Clinical Cardiology Council, Cardiovascular Radiology and Intervention Council, and the Atherosclerotic Peripheral Vascular Disease and Quality of Care Outcomes in Research Interdisciplinary Working Groups: the American Academy of Neurology affirms the value of this guideline as an educational tool for neurologists. Stroke. 2007 May;38(5):1655-711. doi: 10.1161/STROKEAHA.107.181486. Epub 2007 Apr 12. PMID 17431204
- [Result] Broderick J, Connolly S, Feldmann E, Hanley D, Kase C, Krieger D, Mayberg M, Morgenstern L, Ogilvy CS, Vespa P, Zuccarello M; American Heart Association; American Stroke Association Stroke Council; High Blood Pressure Research Council; Quality of Care and Outcomes in Research Interdisciplinary Working Group. Guidelines for the management of spontaneous intracerebral hemorrhage in adults: 2007 update: a guideline from the American Heart Association/American Stroke Association Stroke Council, High Blood Pressure Research Council, and the Quality of Care and Outcomes in Research Interdisciplinary Working Group. Stroke. 2007 Jun;38(6):2001-23. doi: 10.1161/STROKEAHA.107.183689. Epub 2007 May 3. PMID 17478736
- [Result] de Werra I, Jaccard C, Corradin SB, Chiolero R, Yersin B, Gallati H, Assicot M, Bohuon C, Baumgartner JD, Glauser MP, Heumann D. Cytokines, nitrite/nitrate, soluble tumor necrosis factor receptors, and procalcitonin concentrations: comparisons in patients with septic shock, cardiogenic shock, and bacterial pneumonia. Crit Care Med. 1997 Apr;25(4):607-13. doi: 10.1097/00003246-199704000-00009. PMID 9142024